CLINICAL TRIAL: NCT02546349
Title: The Treatment Effect of Inhaled Corticosteroid and Long-acting beta2 Agonist Combination Versus Long-acting Anti-cholinergic Agent on Stratified COPD Patients Based on the Levels of Exhaled Nitric Oxide
Brief Title: Exhaled NO Based Treatment of Chronic Obstructive Pulmonary Disease (COPD), ICS/LABA Versus LAMA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140420
Record Dates: First submitted 2015-02-25; First posted 2015-09-10 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: COPD
Keywords: chronic obstructive pulmonary disease; airway inflammation; eosinophilic airway inflammation; exhaled nitric oxide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone; Salmeterol Xinafoate; Tiotropium Bromide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- high eNO: ICS/LABA (Experimental): patients with eNO >=23.5 ppb, receive inhaled corticosteroid (ICS)/long-acting beta2 agonist (ICS/LABA) of fluticasone/salmeterol 250/25 mcg/puff, 2 puffs bid.
  Interventions: Drug: fluticasone/salmeterol, tiotropium
- high eNO: LAMA (Active Comparator): patients with eNO >=23.5 ppb, receive long acting muscarinic antagonist (LAMA) of tiotropium 2 inhalations 2.5 mcg/inhalation, once daily
  Interventions: Drug: fluticasone/salmeterol, tiotropium
- Low eNO: ICS/LABA (Experimental): patients with eNO < 23.5 ppb, receive fluticasone/salmeterol 250/25 mcg/puff, 2 puffs bid
  Interventions: Drug: fluticasone/salmeterol, tiotropium
- Low eNO: LAMA (Active Comparator): patients with eNO < 23.5 ppb, receive tiotropium 2 inhalations 2.5 mcg/inhalation, once daily
  Interventions: Drug: fluticasone/salmeterol, tiotropium

INTERVENTIONS:
Drug: fluticasone/salmeterol, tiotropium — In group (either high or low eNO), patients will be randomized to receive either 2 puffs of fluticasone/salmeterol 250/25 mcg/puff twice daily or 2 inhalations of tiotropium respimat 2.5 mcg/inhalation once daily for 12 weeks.
  Other Names: seretide evohaler 250; spiriva respimat

SUMMARY:
It is recognized that eosinophilic airway inflammation is more likely respond to steroid treatment. However, in real-world practice, it is difficult to routinely assess airway inflammation using sputum induction because of technical and facility requirement. COPD (chronic obstructive pulmonary disease) is a heterogeneous disease and it remains a great challenge to identify patients who have eosinophilic airway inflammation and respond to steroid treatment well. A recent study demonstrated elevated plasma D-dimer was associated with acute inflammation and a significant predictor of pulmonary embolism in COPD exacerbated patients. D-dimer may potentially act as a marker of inflammation and a predictor of cardiovascular event in COPD patients. The investigators preliminary study demonstrated that exhaled nitric oxide (eNO) > 23.5 ppb is a good surrogate marker to predict eosinophilic airway inflammation in COPD patients who were newly diagnosed or untreated for at least 3 months. There were significant correlations among sputum eosinophils, eNO and serum total immunoglobulin E (IgE). Particularly, eNO predicted sputum eosinophilia (> 3%) in COPD at a sensitivity and specificity of 62% and 71% respectively. Herein, the investigators test the hypothesis that eNO may act as a biomarker to determine treatment option for COPD.

DETAILED DESCRIPTION:
Eligible COPD patients (newly diagnosed or untreated for at least 3 months) will be enrolled at out-patient clinic after consenting by participants. Upon enrollment, exhaled NO (eNO) will be measured and patients will be categorized into 2 groups according to eNO levels: either high exhaled NO (greater than or equal to 23.5 ppb) or low eNO (< 23.5 ppb) group. In each group, patients will be randomized to receive either 2 inhalations of fluticasone/salmeterol 250/25 mcg/ pudd twice daily or 2 inhalations of tiotropium 2.5 mcg/inhalation for 12 weeks and followed at scheduled visits. Testing outcome measures include eNO, lung function, different count and mediators in induced sputum, and which will be tested as the following timings: before (baseline, week 0), and after treatment (week 4 and week 12). Rescue medication and drug compliance will be record.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients aged from 40 to 90 years
2. Current or ex-smoker, with smoking history ≧ 20 pack- years
3. Newly diagnosed or untreated (at least 3 months) COPD patients (forced expiratory volume in first second (FEV1)/forced vital capacity (FVC) < 70%) with post-bronchodilator FEV1 < 80 % predicted value.

Exclusion Criteria:

1. Concurrent allergic rhinitis, eczema, and asthma.
2. Clinically overt bronchiectasis, lung cancer, active tuberculosis, or other known specific pulmonary disease.
3. A chest X-ray indicating diagnosis other than COPD that might interfere with the study.
4. Major disease abnormalities are uncontrolled on therapy.
5. Alcohol or medication abuse.
6. Patients had lower respiratory tract infections or received systemic steroid in the 4 weeks prior to the commencement of study.
7. Women with childbearing potential during the period of trial.
8. Unable or unwilling to comply with all protocol

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Changes of eNO level | Changes of eNO level (ppb) from baseline at 12 weeks

SECONDARY OUTCOMES:
Changes of lung function parameters (FEV1, FVC) | Changes of lung function parameters (FEV1, FVC) from baseline at 12 weeks
Changes of serum level of IgE | Changes of serum level of IgE (IU/ml) from baseline at 12 weeks
Changes of serum level of matrix metalloproteinase (MMP)-9 | Changes of serum level of MMP-9 (ng/ml) from baseline at 12 weeks
Changes of serum level of D-dimer | Changes of serum level of D-dimer (ug/ml) from baseline at 12 weeks
Changes of scales of life quality questionnaire | Changes of scales of life quality questionnaire from baseline at 12 weeks
  COPD assessment test (CAT)
Changes of proportion of cell counts in induced sputum | Changes of proportion of cell counts in induced sputum from baseline at 12 weeks
Changes of MMP-9 level in induced sputum | Changes of MMP-9 levle (ug/ml) in induced sputum from baseline at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diahn-Warng S Perng, PhD, Study Chair — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Derived] Su KC, Ko HK, Hsiao YH, Chou KT, Chen YW, Yu WK, Pan SW, Feng JY, Perng DW. Fractional Exhaled Nitric Oxide Guided-Therapy in Chronic Obstructive Pulmonary Disease: A Stratified, Randomized, Controlled Trial. Arch Bronconeumol. 2022 Aug;58(8):601-610. doi: 10.1016/j.arbres.2021.11.013. Epub 2021 Dec 18. English, Spanish. PMID 35312525